CLINICAL TRIAL: NCT06523465
Title: A Prospective, Multi-center, Randomized Trial to Compare Statin Combined with CCB to MRA Combined with CCB in Primary Aldosteronism Treatment
Brief Title: Statin Combined with Amlodipine Treats Primary Aldosteronism
Acronym: STOP-PA
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Third Military Medical University (Other)
Responsible Party: Principal Investigator, Zhiming Zhu, Department of Hypertension and Endocrinology, Third Military Medical University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: STOP-PA
Record Dates: First submitted 2024-07-17; First posted 2024-07-26 (Actual); Last update posted 2024-11-22 (Actual); Status verified 2024-11

CONDITIONS: Primary Aldosteronism; Statin; Mineralocorticoid Receptor Antagonist; Hypertension
Keywords: primary aldosteronism; hypertension; Statin
MeSH Terms: conditions — Hyperaldosteronism; Hypertension | interventions — Amlodipine; Spironolactone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Simvastatin combined with Amlodipine besylate (Experimental): after 1:1 randomization, 60 patients with primary aldosteronism were treated with Simvastatin combined with Amlodipine besylate for 6 months
  Interventions: Drug: Simvastatin combined with Amlodipine besylate
- Simvastatin combined with Spironolactone and Amlodipine besylate. (Experimental): after 1:1 randomization, 60 patients with primary aldosteronism were treated with Simvastatin combined with Spironolactone and Amlodipine besylate for 6 months
  Interventions: Drug: Simvastatin combined with Spironolactone and Amlodipine besylate.
- Amlodipine besylate combined with Spironolactone (Experimental): after 1:1 randomization, 60 patients with primary aldosteronism were treated with Amlodipine besylate combined with Spironolactone for 6 months
  Interventions: Drug: Amlodipine besylate combined Spironolactone

INTERVENTIONS:
Drug: Simvastatin combined with Amlodipine besylate — 6-month treatment of Simvastatin combined with Amlodipine besylate
  Arms: Simvastatin combined with Amlodipine besylate
Drug: Simvastatin combined with Spironolactone and Amlodipine besylate. — 6-month treatment of Simvastatin combined with Spironolactone and Amlodipine besylate.
  Arms: Simvastatin combined with Spironolactone and Amlodipine besylate.
Drug: Amlodipine besylate combined Spironolactone — 6-month treatment of Amlodipine besylate combined with Spironolactone
  Arms: Amlodipine besylate combined with Spironolactone

SUMMARY:
The drug treatment for primary aldosteronism (PA) is limited and difficult to improve long-term cardiovascular outcomes. This study plans to enroll patients with primary aldosteronism and randomly divide into 3 groups: scheme 1: Statin combined with amlodipine besylate, scheme 2: Statin combined with Spironolactone and Amlodipine besylate. scheme 3: Amlodipine besylate combined with Spironolactone , to observe the changes in plasma aldosterone level, 24-hour urinary aldosterone, blood pressure, and long-term cardiovascular risk.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of primary aldosteronism

Exclusion Criteria:

* Allergy to drugs in this study
* Pregnancy
* Severe liver and kidney dysfunction
* Mental illness

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 180 (Estimated)
Dates: Start 2024-09-10 (Actual); Primary Completion 2025-12-30 (Estimated); Study Completion 2026-09-30 (Estimated)

PRIMARY OUTCOMES:
changes in plasma aldosterone levels | 6 month
  blood samples are collected at baseline and 6 months after treatment to measure plasma aldosterone levels， and compare between groups and within groups (pg/ml)
changes in 24-hour urinary aldosterone levels | 6 month
  24 hours urine are collected at baseline and 6 months after treatment to measure 24-hour urinary aldosterone， and compare between groups and within groups(pmol/24h)

SECONDARY OUTCOMES:
changes in office blood pressure and home blood pressure | 6 month
  Record office blood pressure at baseline and at follow-up after medical treatment (mmHg), and compare between groups and within groups
changes in serum potassium levels | 6 month
  blood samples are collected at baseline and 6 months after treatment to measure serum potassium levels， and compare between groups and within groups (mmol/L)
changes in serum renin level | 6 month
  blood samples are collected at baseline and 6 months after treatment to measure serum renin levels, and compare between groups and within groups (mU/L)
changes in plasma cholesterol levels | 6 month
  blood samples are collected at baseline and 6 months after treatment to measure plasma cholesterol levels， and compare between groups and within groups (mmol/L)
changes in blood glucose | 6 month
  blood samples are collected at baseline and 6 months after treatment to measure blood glucose， and compare between groups and within groups (mmol/L)

CONTACTS AND LOCATIONS:
Locations (1):
- No. 10 Changjiang River Branch, Yuzhong District，Chongqing, China, Chongqing, Chongqing Municipality, China

IPD SHARING:
Plan to Share IPD: No